CLINICAL TRIAL: NCT06680336
Title: Cognitive Recovery After Post Stroke Delirium [RECOVER] a Longitudinal Pilot Proof of Concept Study in Stroke Patients With/without Delirium
Brief Title: Cognitive Recovery After Post Stroke Delirium (RECOVER)
Acronym: RECOVER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AKF_1004-0-0
Record Dates: First submitted 2024-07-08; First posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-07

CONDITIONS: Post Stroke Delirium; Cognitive Functioning After Stroke

STUDY DESIGN:
Intervention Model Description: Longitudinal study with 3 measurements (S1, S2, S3) and two groups of stroke patients (post-stroke-delirium (PSD) patients, non PSD patients)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Post-stroke Delirium (Other): Assessment of cognitive functioning using a multi-component neuropsychological assessment and tasked-based functional MRI (introducing a modified working memory task) at three time points S1, S2, S3.
  Interventions: Diagnostic Test: Mulit-componant neuropsychological assessment; Diagnostic Test: Multimodal MRI
- Non-post-stroke Delirium (Other): Assessment of cognitive functioning using a multi-component neuropsychological assessment and tasked-based functional MRI (introducing a modified working memory task) at three time points S1, S2, S3.
  Interventions: Diagnostic Test: Mulit-componant neuropsychological assessment; Diagnostic Test: Multimodal MRI

INTERVENTIONS:
Diagnostic Test: Mulit-componant neuropsychological assessment — Multi-component cognitive assessment including following domains: attention & information speed, executive functioning, verbal memory, language, visuospatial-construction and orientation.
Diagnostic Test: Multimodal MRI — Structural MRI (e.g., MPRAGE, DTI) and functional MRI (introducing a modified working memory task for stroke patients)

SUMMARY:
RECOVER is a Proof-of-Concept study on cognitive functioning following a longitudinal design with three measurements (during the acute- and post-acute phases of a stroke and a 3-month follow-up) and two equally-sized stroke patient groups: a post-stroke delirium(PSD), and a non-PSD group (control group). Cognitive functioning will be assessed using a multi-component neuropsychological assessment and tasked-based functional MRI (introducing a modified working memory task).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 years
* Ischemic stroke: Stroke Onset ≤ 96h, hospital admission ≤ 48h
* NIHSS ≥ 1
* Informed consent by patient or legal guardian

Exclusion Criteria:

* Aphasia
* Pre-existing conditions such as Dementia, psychiatric disorders (e.g., Depression, Schizophrenia)
* MRI contraindication such as certain metal implants
* Reduced consciousness, defined as Glasgow Coma Scale (GCS) ≤ 8
* Delirium onset before study enrollment

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Global post-stroke cognitive functioning | 90 days
  The primary endpoint will be a between-group comparison of the cognitive outcome, defined as global post-stroke cognitive functioning, at 3 months follow-up (S3), using multimodal data generated from the neuropsychological assessment and tasked-based fMRI.

SECONDARY OUTCOMES:
Domain specific post-stroke cognitive functioning | 90 days
  The second endpoint will be a between-group comparison of the cognitive outcome, defined as domain specific post-stroke cognitive functioning, at 3 months follow-up, using multimodal data generated from the neuropsychological assessment and tasked-based fMRI.
Prediction of global post-stroke cognitive outcome | 5 - 90 days
  A multivariate linear regression model will be used to establish a multi-item prognostic or predictive tool for cognitive outcome, defined as global post-stroke cognitive functioning at the follow-up measurement (S3) by parameters assessed at S1.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology, University Hospital Tuebingen, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No